CLINICAL TRIAL: NCT04580459
Title: Connecting and Reflecting Experience (CARE) Mentalizing-Focused Parenting Group Treatment Outcomes Study
Brief Title: CARE Mentalizing-Focused Parenting Group Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: The FAR Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11240
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Parent-Child Relationship; Parenting
Keywords: Attachment; Parenting; Parent-Child Relationship; Caregivers; Parents; Child Mental Health; Child Development
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARE Parenting Group Treatment (Experimental): Participants receive the CARE mentalizing-focused group parenting intervention.
  Interventions: Behavioral: CARE Parenting Group Treatment
- Treatment as Usual (TAU) (Other): Participants continue to receive treatment as usual in the outpatient child mental health clinic.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: CARE Parenting Group Treatment — The CARE parenting group treatment is a 12-session, 60-minute group mentalizing-focused intervention with 3 monthly parent-child sessions.
  Arms: CARE Parenting Group Treatment
Behavioral: Treatment as Usual (TAU) — Treatment as usual (TAU) involves typical child outpatient mental health services, such as individual child appointments and medication management.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The primary objective of this clinical trial is to evaluate the 12-week mentalizing-focused group parenting intervention, Connecting and Reflecting Experience (CARE), relative to a treatment as usual (TAU) group in an outpatient child mental health clinic.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of child receiving mental health services at community child outpatient clinic
* English- or Spanish-speaking

Exclusion Criteria:

* Parent has severe mental illness or significant cognitive impairment
* Child has significant developmental delay

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in parental reflective functioning | Baseline to post-intervention (12 weeks)
  Change in parental reflective functioning as measured by parent/caregiver report on the Parental Reflective Functioning Questionnaire. Responses are reported on a 7-point Likert scale from 1 to 7. Total scores for the three sub-scales (Pre-Mentalizing Modes, Certainty about Mental States, and Interest and Curiosity) range from 6 to 42. Lower scores on Pre-Mentalizing Modes, moderate scores on Certainty about Mental States, and higher scores on Interest and Curiosity indicate better outcomes.
Change in parenting stress | Baseline to post-intervention (12 weeks)
  Change in parenting stress as measured by parent/caregiver report on the Parenting Stress Index. Responses are reported on a 5-point Likert scale from 1 to 5. Total scores for the Parenting Stress Index (PSI-SF-4) range from 36 to 180, with lower scores indicating better outcomes.

SECONDARY OUTCOMES:
Change in parent psychiatric distress | Baseline to post-intervention (12 weeks)
  Change in parent/caregiver psychiatric distress as measured by parent/caregiver report on the Brief Symptom Inventory. Responses are reported on a 5-point Likert scale from 0 to 4. Global severity index scores for the Brief Symptom Inventory (BSI-18) range from 0 to 82, with lower scores indicating better outcomes.
Change in child social-emotional impairment | Baseline to post-intervention (12 weeks)
  Change in children's social-emotional impairment as measured by parent/caregiver and child report on the Youth Outcome Questionnaire. Responses are reported on a 5-point Likert scale from 0 to 4. Total scores on the Youth Outcomes Questionnaire (Y-OQ-30.2) range from 0 to 120, with lower scores indicating better outcomes.
Change in family functioning | Baseline to post-intervention (12 weeks)
  Change in family functioning as measured by parent/caregiver and child report on the Family Assessment Device. Responses are reported on a 4-point Likert scale from 1 to 4. Total scores on the General Functioning scale of the Family Assessment Device range from 12 to 48, with lower scores indicating better outcomes.
Change in parent emotion regulation | Baseline to post-intervention (12 weeks)
  Change in parent/caregiver emotion regulation as measured by parent/caregiver report on the Difficulties with Emotion Regulation Scale. Responses are reported on a 5-point Likert scale from 1 to 5. Total scores for the Difficulties with Emotion Regulation Scale (DERS-18) range from 18 to 90, with lower scores indicating better outcomes.
Change in parent perceptions of social support | Baseline to post-intervention (12 weeks)
  Change in parent/caregiver perceptions of social support as measured by parent/caregiver report on the Interpersonal Support Evaluation List. Responses are reported on a 4-point Likert scale from 0 to 3. Total scores on the Interpersonal Support Evaluation List (ISEL-12) range from 0 to 36, with higher scores indicating better outcomes.
Change in parent perceptions of belongingness | Baseline to post-intervention (12 weeks)
  Change in parent/caregiver perceptions of belongingness as measured by parent/caregiver report on the Sense of Belongingness Inventory. Responses are reported on a 4-point Likert scale from 1 to 4. Total scores for the Psychological Experience scale of the Sense of Belongingness Inventory range from 18 to 72, with higher scores indicating better outcomes.
Change in parent-child relationship | Baseline to post-intervention (12 weeks)
  Change in parent-child relationship as measured by child report on the Security Scale. Responses are reported on a 4-point Likert scale from 1 to 4. Total scores on the Security Scale range from 1 to 96, with higher scores indicating better outcomes.
Change in reported exposure to adverse childhood experiences (ACEs) | Baseline and post-intervention (12 weeks)
  Change in reported parent and child exposure to ACEs as measured by parent/caregiver report on the Adverse Childhood Experiences (ACE) questionnaire. Responses are reported on a binary (yes/no) scale. Total scores on the Adverse Childhood Experiences questionnaire range from 0 to 10.
Change in parent experiences of racism and discrimination | Baseline and post-intervention (12 weeks)
  Change in reported distress in relation to experiences of racism and/or discrimination as measured by parent/caregiver report on the Daily Life Experiences scale of the Racism and Life Experience Scales. Responses are reported on two 6-point Likert scales from 0 to 5. Total scores on the Daily Life Experiences scale of the Racism and Life Experience Scales range from 0 to 100, with lower scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Zayde, PsyD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zayde A, Derella OJ, Kilbride A. Safe haven in adolescence: Improving parental reflective functioning and youth attachment and mental health with the Connecting and Reflecting Experience. Infant Ment Health J. 2023 Mar;44(2):268-283. doi: 10.1002/imhj.22042. Epub 2023 Mar 2. PMID 36862314